CLINICAL TRIAL: NCT02304536
Title: Comparison Between Laproscopic Ovarian Diathermy and Urinary Purified FSH in Women With Clomiphene Citrate Resistant Polycystic Ovarian Syndrome: A Randomised Controlled Trial
Brief Title: Comparison Between Laparoscopic Ovarian Diathermy and Urinary Purified FSH in Women With Clomiphene Citrate Resistant Polycystic Ovarian Syndrome.
Acronym: FSH
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, AbdelGany Hassan, Lecturer of Gynecology and Obstetrics, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Sub5
Record Dates: First submitted 2014-11-25; First posted 2014-12-02 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FSH (Active Comparator): will receive urinary purified FSH (Fostimon® IBSA, Switzerland) 75IU daily for 7 days starting from the 3rd day of menstruation or progesterone withdrawal bleeding. If the follicle does not exceed 9mm the dose will be increased by 37.5IU every 7 days. The cycle will be cancelled if no follicles exceed 9mm 4 weeks after starting FSH. This was combined with oral metformin (Cidophage® CID, Egypt) 500 mg three times per day.
  Interventions: Drug: FSH
- Ovarian drilling (Active Comparator): 70 women will have laparoscopic ovarian drilling in which the ovaries will be stabilised by grasping the ovarian ligament and monopolar diathermy will be used to do 4-10 punctures in each ovary. The number of punctures will be individualised according to the size of the ovary. Serial vaginal ultrasound scans were done starting from the 10th day of menstruation, the frequency of monitoring will be individualized according to the women's response.
  Interventions: Procedure: Laparoscopic ovarian drilling

INTERVENTIONS:
Drug: FSH — 70 women will receive urinary purified FSH (Fostimon® IBSA, Switzerland) 75IU daily for 7 days starting from the 3rd day of menstruation or progesterone withdrawal bleeding. If the follicle does not exceed 9mm the dose will be increased by 37.5IU every 7 days. The cycle will be cancelled if no follicles exceed 9mm 4 weeks after starting FSH. This was combined with oral metformin (Cidophage® CID, Egypt) 500 mg three times per day
  Arms: FSH
Procedure: Laparoscopic ovarian drilling — 70 women will have LOD in which the ovaries will be stabilised by grasping the ovarian ligament and monopolar diathermy will be used to do 4-10 punctures in each ovary. The number of punctures will be individualised according to the size of the ovary. Serial vaginal ultrasound scans were done starting from the 10th day of menstruation, the frequency of monitoring will be individualized according to the women's response.
  Arms: Ovarian drilling

SUMMARY:
210 women with clomiphene resistant PCOS will be randomly divided into 3 equal groups using computer generated random numbers. Group 1 will receive combined metformin and FSH, group 2 will have LOD and group 3 will act as the control group with no intervention.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is the most common endocrine disorder in reproductive age, with an incidence of 5 -10% . Classically clomiphene citrate (CC) is the first approach to induce ovulation in patients with PCOS. Although 70-80% of PCOS women can ovulate by the treatment with CC, only 40%of the PCOS women become pregnant. Women who do not ovulate with increasing doses of CC are described as being CC-resistant and remain a major challenge in gynecologic endocrinology. Traditional alternatives for CC-resistant patients include gonadotropin therapy and laparoscopic ovarian diathermy.

Gonadotropin therapy is widely used for ovulation induction in CC-resistant PCOS patients. The use of purified FSH preparation virtually free of LH activity, is a recommendable treatment since there is evidence that pure FSH may significantly reduce tonic LH levels, favourably alter the intraovarian hormonal milieu, and promote the initial follicular development with minimal risk of multiple follicular growth or ovarian hyperstimulation .

The use of metformin in PCOS is associated with cycle regulation, improved ovulation, and a reduction in circulating androgen levels (5). Metformin likely plays its role in improving ovulation induction in women with PCOS through a variety of actions, including reducing insulin levels and altering the effect of insulin on ovarian androgen biosynthesis, theca cell proliferation, and endometrial growth. In addition, potentially through a direct effect, it inhibits ovarian gluconeogenesis and thus reduces ovarian androgen production .

Laparoscopic ovarian drilling (LOD) can avoid or reduce the need for gonadotropins for ovulation induction. Several potential mechanisms of action of LOD have also been suggested. The reduction of inhibin production following LOD is followed by an increase in FSH secretion and recruitment of a new cohort of follicles. Other theory is restoration of normal production of the putative gonadotropin surge after laparoscopic ovarian electrocautery. Moreover, drainage of androgens and inhibin from follicles surface may inhibit the excessive collagenisation of overlying ovarian cortex and facilitate Softening of ovarian tunica. Neighbouring follicles that are not undergoing atresia may then mature and gain access to the ovarian surface, facilitating ovulation. Initiation of normal inhibin B pulsatility by LOD appears to correlate with the postoperative onset of ovulatory cycles (3).

The main drawbacks of LOD are adhesions formation and ovarian atrophy. That is why minimising the number of diathermy points and avoiding diathermy near the ovarian hilum are recommended.

All women with clomiphene resistant PCOS attending the subfertility clinic of Cairo university hospitals will be invited to participate in the study. PCOS diagnosis will be based on chronic anovulation and sonographic picture of polycystic ovaries (8). Clomiphene resistance will be defined as failure of ovulation in spite of receiving 150mg of clomiphene citrate for 5 days during the menstrual cycle.

Exclusion criteria are age >40 years, other causes of infertility, hyperprolactinaemia, allergy to FSH or metformin, previous FSH or LOD therapy, and body mass index (BMI)>35.

The study will be explained to all the participants and a written informed consent will be obtained before participation.

Full history will be taken followed by complete examination and sonographic evaluation. Sonographic picture of polycystic ovaries will be defined when there are at least 12 follicles 2-9mm in the ovary and/or ovarian volume>10cm3.

210 women with clomiphene resistant PCOS will be randomly divided into 3 equal groups using computer generated random numbers. Group 1 will receive combined metformin and FSH, group 2 will have LOD and group 3 will act as the control group with no intervention.

Group 1 will receive urinary purified FSH (Fostimon® IBSA, Switzerland) 75IU daily for 7 days starting from the 3rd day of menstruation or progesterone withdrawal bleeding. If the follicle does not exceed 9mm the dose will be increased by 37.5IU every 7 days. The cycle will be cancelled if no follicles exceed 9mm 4 weeks after starting FSH. This was combined with oral metformin (Cidophage® CID, Egypt) 500 mg tds.

Group 2 will have LOD in which the ovaries will be stabilised by grasping the ovarian ligament and monopolar diathermy will be used to do 4-10 punctures in each ovary. The number of punctures will be individualised according to the size of the ovary. Serial vaginal ultrasound scans were done starting from the 10th day of menstruation, the frequency of monitoring will be individualized according to the women's response.

When the dominant follicle reaches 17mm or more in either group, women will receive Human chorionic gonadotrophin (Choriomon® IBSA, Switzerland) 5000IU and a timed intercourse will be advised 36 hours later.

Group 3 will have regular progesterone withdrawal bleeding in the form of norethisterone (stereonate® Hi Pharm, Egypt).

ELIGIBILITY:
Inclusion Criteria:

* Clomiphene resistant PCOS

Exclusion Criteria:

* Other causes of infertility
* Hyperprolactinaemia.
* Allergy to FSH.
* BMI>35

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 210 (Estimated)
Dates: Start 2014-11; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Ovulation | 6 weeks after starting the intervention
  Vaginal sonography will be done regularly to check ovulation.

SECONDARY OUTCOMES:
Proportion of women getting pregnant | 6 months after starting the intervention
  Pregnancy will be diagnosed by the presence of an intrauterine gestational sac on vaginal ultrasound scan one week after a missed period.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - BeniSuef University hospitals, BeniSuef
  - Cairo University Hospitals, Cairo

REFERENCES:
- [Background] van Wely M, Bayram N, van der Veen F, Bossuyt PM. Predictors for treatment failure after laparoscopic electrocautery of the ovaries in women with clomiphene citrate resistant polycystic ovary syndrome. Hum Reprod. 2005 Apr;20(4):900-5. doi: 10.1093/humrep/deh712. Epub 2005 Jan 7. PMID 15640254
- [Background] Sam S, Dunaif A. Polycystic ovary syndrome: syndrome XX? Trends Endocrinol Metab. 2003 Oct;14(8):365-70. doi: 10.1016/j.tem.2003.08.002. PMID 14516934